CLINICAL TRIAL: NCT03177785
Title: Testing a Resilience Intervention for Individuals Aging With Multiple Sclerosis (MS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Dawn Ehde, Professor, Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 47142
Record Dates: First submitted 2017-04-03; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Intervention (Experimental): 6-weeks of telephone-delivered sessions, moderated by a trained clinician offering EverydayMatters MS.
  Interventions: Behavioral: EverydayMatters
- Control (No Intervention): Wait-list control

INTERVENTIONS:
Behavioral: EverydayMatters
  Arms: Intervention

SUMMARY:
This study aims to test the efficacy of the EverydayMatters Multiple Sclerosis (MS) program for individuals age 45 or older living with multiple sclerosis. The program involves a 6-week telephone-delivered program to promote resilience and happiness for individuals living with MS.

ELIGIBILITY:
Inclusion Criteria:

* 45 years of age
* Diagnosis of multiple sclerosis
* regular access to the phone and internet
* willing to join a moderated group on MSConnection.org

Exclusion Criteria:

* under 45 years of age
* no diagnosis of multiple sclerosis
* no access to the phone or internet
* unwilling to join moderated group on MSConnection

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Resilience using Connor Davidson Resilience Scale (brief) | 6 weeks
  10-item self-report measure of resilience.

SECONDARY OUTCOMES:
Change in positive affect and well being using the Quality of Life in Neurological Disorders (NeuroQoL) Positive Affect and Well-Being Short Form | 6 weeks
  9-item self report measure
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Satisfaction with Social Roles Short Form | 6 weeks
  4-item self-reported measure of satisfaction with participation in social roles and activities
Change in disease-management self-efficacy using the University of Washington Self-Efficacy Scale | 6 weeks
  6-item self-report measure of self-efficacy for disability management

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Ehde, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alschuler KN, Arewasikporn A, Nelson IK, Molton IR, Ehde DM. Promoting resilience in individuals aging with multiple sclerosis: Results from a pilot randomized controlled trial. Rehabil Psychol. 2018 Aug;63(3):338-348. doi: 10.1037/rep0000223. Epub 2018 Jul 19. PMID 30024203